CLINICAL TRIAL: NCT05934968
Title: The Effects of the 6-week Mad Dog Anti-inflammatory Cooking Class Series on Dietary Self-efficacy, Eating Behaviors and Health Outcomes in People With Neurological Disability
Brief Title: Mad Dog Cooking Class Series: Effects on Dietary Self-efficacy, Eating Behaviors and Health Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, David Ditor, Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-337 - Ditor
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis; Diet, Healthy; Inflammation; Depression; Adherence, Treatment
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Inflammation; Depression; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mad Dog cooking class intervention group (Experimental): This 6-week series consists of a once-weekly cooking class and educational session where a group of individuals with neuromuscular disability can come together to learn about the health benefits of an anti-inflammatory diet, receive instruction on how to cook selected anti-inflammatory recipes, and experiment with various pieces of accessible kitchen equipment that may increase their meal preparation skills. This series will also allow participants to share a meal together once per week.
  Interventions: Other: Mad Dog cooking class series
- Control group (No Intervention): The control group will be given the Mad Dog recipes but will not take part in the Mad Dog cooking class series.

INTERVENTIONS:
Other: Mad Dog cooking class series — This 6-week series consists of a once-weekly cooking class and educational session where a group of individuals with neuromuscular disability can come together to learn about the health benefits of an anti-inflammatory diet, receive instruction on how to cook selected anti-inflammatory recipes, and experiment with various pieces of accessible kitchen equipment that may increase their meal preparation skills. This series will also allow participants to share a meal together once per week.
  Arms: Mad Dog cooking class intervention group

SUMMARY:
Spinal cord injury (SCI) and multiple sclerosis (MS) are both conditions characterized by chronic inflammation as indicated by elevated levels of circulating pro-inflammatory cytokines. These cytokines can have a wide array of negative impacts such as increasing the risk of depression and the intensity and frequency of neuropathic pain.

Recent work in the investigator's laboratory has shown that a 3-month anti-inflammatory diet is not only effective in reducing pro-inflammatory cytokines, but also in reducing depression and neuropathic pain, by approximately 55% and 40%, respectively. However, a one-year follow-up study from the investigator's lab showed such adherence to be very challenging and therefore, strategies are required to address barriers to healthy eating in those with neurological disability.

Accordingly, the investigators have developed a modified anti-inflammatory diet (Mad Dog diet) that is more palatable, less expensive and less demanding, as well as a 2-part pre-diet consultation that effectively increased self-efficacy for dietary adherence, and actual adherence one month post-consult. Still, participant feedback suggests that further efforts are needed to help ensure long term adherence to anti-inflammatory diets for those with neurological disability.

As such, the investigators have developed the 6-week Mad Dog cooking series. This series consists of a once-weekly cooking class and educational session where a group of individuals with neuromuscular disability can come together to learn about the health benefits of an anti-inflammatory diet, receive instruction on how to cook selected anti-inflammatory recipes, and experiment with various pieces of accessible kitchen equipment that may increase their meal preparation skills.

The purpose of this study is to test the 6-week Mad Dog cooking series in individuals with neuromuscular disability to gauge consumer satisfaction and make preliminary measures on self-efficacy for adhering to the Mad Dog anti-inflammatory diet, as well as actual adherence 6 months after the series has been completed. The investigators will also determine if the series has any effect on depressive symptoms.

DETAILED DESCRIPTION:
As mentioned above, the Mad Dog cooking series consists of 6 once-weekly cooking classes and educational sessions where a group of individuals with neuromuscular disability can come together to learn about the health benefits of an anti-inflammatory diet, receive instruction on how to cook selected anti-inflammatory recipes, and experiment with various pieces of accessible kitchen equipment that may increase their meal preparation skills. These classes will take place in the kitchen in the Brock Research and Innovation Centre (130 Lockhart Drive) which is a completely accessible building. The classes will be led by a Brock University graduate student and take approximately 90 minutes each, and each class will have a different theme (See below). This series will also allow participants to share a meal together once per week which the investigators expect (based on past feedback) to foster a sense of community and belonging, improve mood and increase the likelihood of long term adherence to the anti-inflammatory diet.

Schedule:

Week 1: Introduction to Anti-Inflammatory Eating (Veggies and Pita with Mad Dog Hummus, Mad Dog Thai Curry, Mad Dog Nut Mix) Week 2: Focus on Breakfast (Chocolate Protein Smoothie, Poached Eggs Potato Hash and Wilted Kale, Overnight Oats) Week 3: Healthy Flavors of the Globe (Baked Plantain and Sweet Potato Chips, Lentil Tacos with rice and beans, Sugarless Sticky Toffee Pudding) Week 4: Tribute to Canada (Split Pea Soup, Chicken Tourtière with roasted veggies, Nanaimo Bars) Week 5: Anti-Inflammatory Powerhouses (Green Juice, Chicken Breast with Kale and Wild Rice Salad, Turmeric Coconut Bites) Week 6: Protein Positive (White Bean Dip with veggies and crackers, Vegetarian Chili, Sweet Potato Protein Pudding)

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, participants are required to be over 18 years of age, fluent in English and at least one year removed from either spinal cord injury (SCI) or diagnosis of multiple sclerosis (MS). Participants with SCI can have any level or severity of injury while participants with MS can have had any type of MS.

Exclusion Criteria:

* Younger than 18
* Not fluent in English
* No SCI or diagnosis of MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Custom-designed task self-efficacy questionnaire | Baseline (for the intervention group and the control group)
  Confidence in one's abilities to adhere to the anti-inflammatory diet. This is a 4-item questionnaire that asks how confident participants are about adhering to the diet for certain amounts of time at certain percentages of adherence. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 4 and the maximum score is 28, and higher scores indicate greater self-efficacy.
Custom-designed task self-efficacy questionnaire | 6-week timepoint (for the intervention group and the control group)
  Confidence in one's abilities to adhere to the anti-inflammatory diet. This is a 4-item questionnaire that asks how confident participants are about adhering to the diet for certain amounts of time at certain percentages of adherence. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 4 and the maximum score is 28, and higher scores indicate greater self-efficacy.
Custom-designed task self-efficacy questionnaire | 6-month follow-up timepoint (for the intervention group and the control group)
  Confidence in one's abilities to adhere to the anti-inflammatory diet. This is a 4-item questionnaire that asks how confident participants are about adhering to the diet for certain amounts of time at certain percentages of adherence. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 4 and the maximum score is 28, and higher scores indicate greater self-efficacy.
Custom-designed barrier self-efficacy questionnaire | Baseline (for the intervention group and the control group)
  Confidence in one's ability to overcome the barriers associated with adhering to anti-inflammatory diet. This is a 5-item questionnaire that asks participants how confident they are about overcoming the barriers associated with adhering to the anti-inflammatory diet. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 5 and the maximum score is 35, and higher scores indicate greater self-efficacy.
Custom-designed barrier self-efficacy questionnaire | 6-week timepoint (for the intervention group and the control group)
  Confidence in one's ability to overcome the barriers associated with adhering to anti-inflammatory diet. This is a 5-item questionnaire that asks participants how confident they are about overcoming the barriers associated with adhering to the anti-inflammatory diet. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 5 and the maximum score is 35, and higher scores indicate greater self-efficacy.
Custom-designed barrier self-efficacy questionnaire | 6-month follow-up timepoint (for the intervention group and the control group)
  Confidence in one's ability to overcome the barriers associated with adhering to anti-inflammatory diet. This is a 5-item questionnaire that asks participants how confident they are about overcoming the barriers associated with adhering to the anti-inflammatory diet. Each item is scored from 1 (not confident at all) to 7 (completely confident). The minimum score is 5 and the maximum score is 35, and higher scores indicate greater self-efficacy.
Adherence to the anti-inflammatory diet | Baseline (for the intervention group and the control group)
  Participants will complete a 7-day food log. Food logs are then analyzed for the number of servings the participant ate that were approved on the anti-inflammatory diet, the number of servings that were not allowed (cheats) and the total servings eaten over the 7 days. Adherence rates are then determined by calculating [(servings allowed/total servings) * 100.
Adherence to the anti-inflammatory diet | 6-week timepoint (for the intervention group and the control group)
  Participants will complete a 7-day food log. Food logs are then analyzed for the number of servings the participant ate that were approved on the anti-inflammatory diet, the number of servings that were not allowed (cheats) and the total servings eaten over the 7 days. Adherence rates are then determined by calculating [(servings allowed/total servings) * 100.
Adherence to the anti-inflammatory diet | 6-month follow-up timepoint (for the intervention group and the control group)
  Participants will complete a 7-day food log. Food logs are then analyzed for the number of servings the participant ate that were approved on the anti-inflammatory diet, the number of servings that were not allowed (cheats) and the total servings eaten over the 7 days. Adherence rates are then determined by calculating [(servings allowed/total servings) * 100.
Custom-designed consumer satisfaction questionnaire | 6-week timepoint (for the intervention group only)
  Consumer satisfaction with the Mad Dog cooking class series will be measured on a custom designed questionnaire containing 10 items scored on a 7-point scale (1 = strongly disagree, 7 = strongly agree; ex: I feel that I learned new and helpful information in the Mad Dog cooking class series). The minimum score on this questionnaire is 10 and the maximum score is 70, with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
Depression as determined by the Centre for Epidemiological Studies depression (CES-D) | Baseline (for the intervention group and the control group)
  Depression as determined by the Centre for Epidemiological Studies depression (CES-D) This is a 20-item questionnaire that asks participants to rate their depressive symptoms over the last 7 days, and each item is scored from 0-3. The minimum score for the questionnaire 0 and the maximum score is 60, with higher scores indicating worse depressive symptomology. Any score above 15 is indicative of clinical depression, but should not be taken as a diagnosis by itself.
Depression as determined by the Centre for Epidemiological Studies depression (CES-D) | 6-week timepoint (for the intervention group and the control group)
  Depression as determined by the Centre for Epidemiological Studies depression (CES-D) This is a 20-item questionnaire that asks participants to rate their depressive symptoms over the last 7 days, and each item is scored from 0-3. The minimum score for the questionnaire 0 and the maximum score is 60, with higher scores indicating worse depressive symptomology. Any score above 15 is indicative of clinical depression, but should not be taken as a diagnosis by itself.
Depression as determined by the Centre for Epidemiological Studies depression (CES-D) | 6-month follow-up timepoint (for the intervention group and the control group)
  Depression as determined by the Centre for Epidemiological Studies depression (CES-D) This is a 20-item questionnaire that asks participants to rate their depressive symptoms over the last 7 days, and each item is scored from 0-3. The minimum score for the questionnaire 0 and the maximum score is 60, with higher scores indicating worse depressive symptomology. Any score above 15 is indicative of clinical depression, but should not be taken as a diagnosis by itself.

CONTACTS AND LOCATIONS:
Overall Officials: David S Ditor, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Available upon reasonable request to the Principal Investigator